CLINICAL TRIAL: NCT01187641
Title: Comparison of the Diagnostic Accuracy of 3D Volume Acquisition MRI With CT in Staging Colonic Cancer
Status: Completed | Type: Observational
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: CCR3370
Record Dates: First submitted 2010-08-23; First posted 2010-08-24 (Estimated); Last update posted 2017-06-20 (Actual); Status verified 2017-06

CONDITIONS: Colon Cancer
Keywords: cancer, colon, MRI scan
MeSH Terms: conditions — Colonic Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- colon cancer: patients undergoing treatment for colon cancer

SUMMARY:
The purpose of this study is to determine whether MRI is more accurate than CT in determining the T stage, N stage, depth of tumour invasion and extra mural venous invasion (EMVI) preoperatively in colon cancer.

DETAILED DESCRIPTION:
The patient will proceed with their usual colon cancer assessment and treatment, including colonoscopy with biopsy and histology and preoperative CT chest abdomen and pelvis. In addition, patients who enroll in the study will have 2 preoperative MRIs of their abdomen and pelvis performed. One of these will be performed on a 1.5T and the other will be performed on a 3.0T MRI scanner. We will use 20mg of IM buscopan to reduce bowel mobility for each scan. A coronal scout scan will be taken to identify the tumour and select the target volume. IV gadolinium (a contrast agent routinely used in MRI scans to help identify different tissues) will be administered, and a 3D VIBE scan (T1 weighted) will be performed of the target volume. The liver will also be imaged at this time to look for liver metastases. A T2 weighted 3D volume acquisition will then be obtained of the target volume containing the tumour (and its lymphatic drainage).

The MRI will be independently reported by an expert without knowledge of the results of any other investigations. The results of the MRI scan will then be made available to the clinical team. The patient will then proceed as normal with any other investigation which the clinical team feel is necessary, and be treated as normal for their colon cancer. The patient will proceed with their surgery as normal, and the specimen removed at the time of the operation will be examined in the pathology laboratory to determine the exact stage of the cancer.

The accuracy of CT and MRI in staging colon cancer will then be determined against the reference standard provided by the histology examination.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing treatment for colon cancer
* patients undergoing primary surgery for colon cancer and who do not require neo-adjuvant therapy on the basis of their pre-operative CT

Exclusion Criteria:

* age <18
* unable to consent
* consent withheld or withdrawn
* Unable to have an MRI (e.g pacemaker, metal implant)
* Allergy or contraindications to busocopam, gadolinium, small bowel contrast agent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with colon cancer
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2010-08-18 (Actual); Primary Completion 2015-03-31 (Actual); Study Completion 2016-05-17 (Actual)

PRIMARY OUTCOMES:
The primary endpoint will be the accuracy of MRI and CT in determining T stage using histology as the gold standard, on a per patient basis.

SECONDARY OUTCOMES:
Secondary endpoints will be the accuracy of CT and MRI in determining N stage, depth of invasion beyond the muscularis propria, and EMVI.
We will also compare the accuracy of 1.5T against 3.0T MRI scans, and T2 weighted against T1 weighted images

CONTACTS AND LOCATIONS:
Overall Officials: Prof Gina Brown, Principal Investigator — Royal Marsden NHS Foundation Trust
Locations (1):
- The Royal Marsden NHS Foundation Trust, Sutton, Surrey, United Kingdom

REFERENCES:
- [Background] Hunter C, Blake H, Jeyadevan N, Abulafi M, Swift I, Toomey P, Brown G. Local staging and assessment of colon cancer with 1.5-T magnetic resonance imaging. Br J Radiol. 2016 Aug;89(1064):20160257. doi: 10.1259/bjr.20160257. Epub 2016 May 26. PMID 27226219
- [Result] Hunter C, Siddiqui M, Georgiou Delisle T, Blake H, Jeyadevan N, Abulafi M, Swift I, Toomey P, Brown G. CT and 3-T MRI accurately identify T3c disease in colon cancer, which strongly predicts disease-free survival. Clin Radiol. 2017 Apr;72(4):307-315. doi: 10.1016/j.crad.2016.11.014. Epub 2017 Jan 31. PMID 28159328